CLINICAL TRIAL: NCT04475718
Title: Fourth Trimester - A Web-based Tool for Postpartum Care to Address the Needs of Underserved Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: Orange Square Design, Inc. (Industry); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Lisa Marceau, Staff Vice President, Digital Research Solutions, Carelon Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R43MD014923 (NIH); R43MD014923 (NIH)
Record Dates: First submitted 2020-07-09; First posted 2020-07-17 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Pregnancy Related; Postpartum Sadness
Keywords: Postpartum health; Fourth trimester; Resiliency; Health disparities; Maternal health; Mobile tools; Human-centered design; Digital health

STUDY DESIGN:
Intervention Model Description: Interviews were conducted with 24 pregnant and postpartum women. From this research and other activities, the investigators built a prototype program. Once the prototype was completed, the investigators conducted a clinical trial with 87 participants. The pre-test captured key outcome measures (resilience, stress, anxiety, depression, fear, knowledge, and variables related to COVID-19) and other descriptive variables. All participants who completed the pre-test were given access to the prototype mobile postpartum tool. Participants were asked to actively engage with the tool for 4 weeks, during which time they provided real-time user experience feedback. At the end of the 4-week period, the investigators conducted a post-test to measure change in outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fourth Trimester Mobile Tool (Other): Fourth Trimester Mobile Tool
  Interventions: Behavioral: Fourth Trimester Mobile Tool

INTERVENTIONS:
Behavioral: Fourth Trimester Mobile Tool — A mobile web-based tool for underserved women in the fourth trimester. The mobile platform teaches self-efficacy, care management, and coping skills to help reduce major health risks and provide tools and resources to maintain mental health.

SUMMARY:
The postpartum period is a critical time for both maternal and child health, and more than half of all maternal deaths occur postpartum, from one day to one year after birth. This poor outcome is linked to the racial and ethnic disparities that disproportionately effects low income and black women. To reduce the burden of the postpartum period for this population, the goal of this project is to develop an accessible, targeted online tool designed to address the needs of underserved women who are at greater risk for adverse postpartum outcomes by providing the appropriate tools, knowledge and skills to improve postpartum health.

DETAILED DESCRIPTION:
In the United States, the postpartum period is a critical time for both maternal and child health, the mortality rate is the highest among other developed, high income countries and more than half of all maternal deaths occur postpartum, from one day to one year after birth. This poor outcome is linked to the racial and ethnic disparities that disproportionately effect black women who are 3-4 times more likely to experience maternal mortality than white women. Recently, the American College of Obstetricians and Gynecologists recognized the deficiencies in postpartum care and coined the term the 'fourth trimester' to mark the time following the birth of the infant through the first 3-months postpartum, and updated its recommendations to address these challenges. With impacts to health outcomes and healthcare costs, there is a need to holistically bridge the gap for low-income and/or ethnically diverse groups of women to address the physical, cultural, and knowledge barriers to accessing quality postpartum care.

To improve the rate at which underserved women are disproportionately affected by maternal mortality and morbidity, the investigators need to engage women leading into and specifically during the postpartum period to identity areas of need, and to provide tools which reduce barriers for women to get appropriate postpartum care. Technology offers innovative solutions to challenges around equal information access. Pregnant women often turn to the internet to find out more information about their health and their developing babies health. Yet, studies find that mothers are not finding sufficient resources to match their postpartum needs.

To address this gap in care, this project aims to develop a mobile tool designed to increase accessibility to information and practical approaches for addressing the complex needs of women in this 'fourth trimester'. This tool will specifically focus on underserved women who are at greatest risk of adverse postpartum outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+;
* Self-reported annual household income less than $39,500 (at least 75% of participants - defined as "low income" household by the PEW Research Center);
* Racial/ethnic minority (at least 75% of participants must be non-white, with at least 50% identifying as Black/African American);
* Be a new or expectant mother - participants must be at least 28 weeks/6 months pregnant (3rd trimester), and up to 6 months post-birth (no more than 10% of participants will be currently pregnant, at least 90% will be postpartum).
* Able to comply with the terms of the study (available time commitment, have internet access; willing to comply with the specified focus groups and survey); and
* Able to read, write and speak English (all research and product development activities will be conducted in English due to budgetary constraints).

Exclusion Criteria:

* Unable to comply with the Inclusion Criteria
* Did not have a live birth (for those who are post-birth)
* Self-reported major medical/health issue which would impact participants' health or ability to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Merz, Principal Investigator — Orange Square Design, Inc.; Lisa Marceau, MPH, Principal Investigator — Carelon Research
Locations (2):
- United States (2):
  - HealthCore, Watertown, Massachusetts
  - Orange Square Design Inc., Pawtucket, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fourth Trimester Mobile Tool
Started | 87
Completed | 79
Not Completed | 8

BASELINE CHARACTERISTICS:
Groups:
- Pre-Post Comparison: Each participant was provided access to the Joyuus prototype for one month. Pilot participants were asked to complete a pretest, answer two real-time experience surveys while using the tool (visual identity and content), and complete a post-test one month after accessing the tool.
Arm/Group | Pre-Post Comparison
Number analyzed (Participants) | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 85
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 79
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 86
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 87

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Resilience at 4 Weeks
Description: Measured by the Connor-Davidson Resilience Scale, a 25-item scale covering 17 domains related to resiliency, used with a variety of populations, across a wide range of languages, racial/ethnic, and cultural groups. It has strong psychometric properties and validated short forms. Scoring of the scale is based on summing the total of all items, each of which is scored from 0-4. For the CD-RISC-25, the full range is from 0 to 100, with higher scores reflecting greater resilience.
Time Frame: baseline, 4 weeks
Population: Analysis of change in outcome between baseline and after one-month will compare change in composite summary scale scores from pre-test to post-test for subjects in the ITT analysis set with data for both time points.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pre-Post Comparison
Number analyzed (Participants) | 87
score on a scale
  Baseline | 26.57 [25.45 to 27.70]
  4 Weeks: number analyzed (Participants) | 79
  4 Weeks | 28.29 [27.11 to 29.45]
  Difference of Post and Pre Total Score for Connor-Davidson Resilience Scale: number analyzed (Participants) | 79
  Difference of Post and Pre Total Score for Connor-Davidson Resilience Scale | 1.85 [.92 to 2.78]
Statistical Analysis 1: Comparison: Pre-Post Comparison; Test type: Other — Preliminary Efficacy; p < .001, t-test, 2 sided

2. Secondary Outcome: Change From Baseline Depressive Symptoms at 4 Weeks Using the Edinburgh Postnatal Depression Scale (EPDS)
Description: The Edinburgh Postnatal Depression Scale (EPDS) will be used to assess depressive symptoms. The 10-question Edinburgh Postnatal Depression Scale (EPDS) is a valuable and efficient way of identifying patients at risk for perinatal depression. Scores range from 0-30. Higher scores indicate more depressive symptoms. Mothers who score above 13 are likely to be suffering from a depressive illness of varying severity.
Time Frame: baseline, 4 weeks
Population: 87 participants completed baseline. 79 participants completed the post-test at 4 weeks.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fourth Trimester Mobile Tool
Number analyzed (Participants) | 87
score on a scale
  Baseline | 8.90 [7.74 to 10.05]
  4 Weeks: number analyzed (Participants) | 79
  4 Weeks | 8.70 [7.56 to 9.83]
  Difference of Post and Pre Total Score for Edinburgh Postnatal Depression Scale: number analyzed (Participants) | 79
  Difference of Post and Pre Total Score for Edinburgh Postnatal Depression Scale | -0.24 [-1.21 to 0.73]

3. Secondary Outcome: Change From Baseline Social Support at 4 Weeks Using the MOS Social Support Survey
Description: The MOS Social Support Survey will be used to assess overall social support and 4 subscales (Emotional/Informational Support; Tangible Support; Affectionate Support; Positive Social Interaction). The MOS Social Support Survey is a 19-item self-administered instrument. Items range from 1-5. The overall social support score is calculated as the mean response to all 19 items. Scores range from 19-95 with higher scores indicating more support.
Time Frame: baseline, 4 weeks
Population: 87 participants completed baseline. 79 participants completed the post-test at 4 weeks.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fourth Trimester Mobile Tool
Number analyzed (Participants) | 87
score on a scale
  Baseline | 3.67 [3.51 to 3.84]
  4 Weeks: number analyzed (Participants) | 79
  4 Weeks | 3.64 [3.45 to 3.84]
  Difference of Post and Pre overall summary score for MOS Social Support: number analyzed (Participants) | 79
  Difference of Post and Pre overall summary score for MOS Social Support | -0.02 [-0.17 to 0.12]

4. Secondary Outcome: Change From Baseline Parent Anxiety at 4 Weeks
Description: The State-Trait Anxiety Inventory (STAI) is a measure of trait and state anxiety with 20 items for assessing trait anxiety and 20 for state anxiety. It has been validated for use with pregnant women. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). The range of possible scores for form Y of the STAI varies from a minimum score of 20 to a maximum score of 80 on both the STAI-T and STAI-S subscales. Higher scores indicate greater anxiety.
Time Frame: baseline, 4 weeks
Population: 87 participants completed baseline. 79 participants completed the post-test at 4 weeks.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pre-Post Comparison
Number analyzed (Participants) | 87
score on a scale
  Baseline | 41.44 [39.38 to 43.49]
  4 Weeks: number analyzed (Participants) | 79
  4 Weeks | 40.87 [38.58 to 43.16]
  Difference of Post and Pre Total score for State-Trait Anxiety Inventory: number analyzed (Participants) | 79
  Difference of Post and Pre Total score for State-Trait Anxiety Inventory | -0.82 [-2.35 to 0.70]

5. Secondary Outcome: Change From COVID-19 and Mental Health Impacts at 4 Weeks
Description: The COVID-19 and Mental Health Impacts tool is a survey to help better understand how the novel coronavirus (COVID-19) pandemic is affecting people's emotional and mental health. A modified version of this instrument was used (removing Q1) to assess the impact of COVID-19 on study participants. All items are rated on a 5-point scale (from Strongly Disagree to Strongly Agree). The range of possible scores is 12-60, with higher scores indicating greater impact of COVID-19. The overall summary score is the sum of all items . While COVID-19 impact was not a formal endpoints, a descriptive analysis of this measure was conducted.
Time Frame: baseline, 4 weeks
Population: 87 participants completed baseline. 79 participants completed the post-test at 4 weeks.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fourth Trimester Mobile Tool
Number analyzed (Participants) | 87
score on a scale
  Baseline | 29.34 [27.34 to 31.35]
  4 Weeks: number analyzed (Participants) | 79
  4 Weeks | 29.65 [27.55 to 31.74]
  Difference of Post and Pre Total score for COVID-19 and Mental Health Impacts: number analyzed (Participants) | 79
  Difference of Post and Pre Total score for COVID-19 and Mental Health Impacts | 0.03 [-1.53 to 1.58]

ADVERSE EVENTS:
Time Frame: AEs were collected for each participant at pre-test and post-test during the four week participation window.
Description: We surveyed participants on health-related measures at two timepoints (pre-test and post-test) and conducted weekly review of participant scores specifically for the Edinburgh Postnatal Depression Scale (EDPS) and the State-Trait Anxiety Inventory (STAI).
  A 0 for all-cause mortality indicates there were no cases of mortality during the study period.
Arm/Group | Fourth Trimester Mobile Tool
All-Cause Mortality (participants affected / at risk) | 0/87
Serious Adverse Events (participants affected / at risk) | 0/87
Other Adverse Events (participants affected / at risk) | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT04475718/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT04475718/SAP_001.pdf